CLINICAL TRIAL: NCT00674752
Title: A Randomized, Double-Blind, Single-Dose, Placebo-Controlled, Multicenter, Polysomnographic Study Of Gabapentin 250 mg And 500 mg In Transient Insomnia Induced By A Sleep Phase Advance
Brief Title: A Polysomnographic Study Of Single-Dose Gabapentin In Transient Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9451157
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2011-04

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Gabapentin
- B (Experimental)
  Interventions: Drug: Gabapentin
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 250 mg oral capsule 30 minutes prior to bedtime
  Arms: A
Drug: Gabapentin — Gabapentin 500 mg oral capsule 30 minutes prior to bedtime
  Arms: B
Drug: Placebo — Matched placebo oral capsule 30 minutes prior to bedtime
  Arms: C

SUMMARY:
The purpose of this study is to assess the effect of gabapentin on polysomnographic assessments in transient insomnia induced by a sleep phase advance.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18 years who reported occasional sleeplessness in the month prior to screening
* Females of child-bearing potential using medically-acceptable method of birth control >/= 1 month prior to screening

Exclusion Criteria:

* Current or recent history (within 2 years) of sleep disorder (excessive snoring, obstructive sleep apnea, chronic painful condition)
* Currently taking or expected to take any of the following during the trial: amphetamines, benzodiazepines, cocaine, marijuana, methaqualone, methadone, opiates, propoxyphene, barbituates, and phencyclidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2006-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Wake after sleep onset as measured by polysomnography (PSG) | Hour +8

SECONDARY OUTCOMES:
PSG Latency to Persistent Sleep | Hour +8
PSG Wake Time During Sleep | Hour +8
PSG WASO | Hour +8
PSG Sleep Onset Latency | Hour +8
Vital signs | Hour +8
Karolinska Sleep Diary-Sleep (KSD) Quality Index | Hour +8
KSD individual scores | Hour +8
PSG NA | Hour +8
Adverse events | Hour +13
PSG Total wake time plus Stage 1 sleep | Hour +8
PSG TST | Hour +8
PSG Sleep Efficiency | Hour +8
PSG Percent of Stages 1, 2, 3, 4 and REM sleep | Hour +8
PSG Percent slow wave sleep (Stages 3&4 combined) | Hour +8
subjective Sleep Latency | Hour +8
subjective Number of Awakenings (NA) | Hour +8
subjective Wake After Sleep Onset (WASO) | Hour +8
subjective Total Sleep Time (TST) | Hour +8
subjective Assessment of Sleep Refreshment | Hour +8
subjective Assessment of Sleep Quality | Hour +8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Cincinnati, Ohio

REFERENCES:
- [Derived] Rosenberg RP, Hull SG, Lankford DA, Mayleben DW, Seiden DJ, Furey SA, Jayawardena S, Roth T. A randomized, double-blind, single-dose, placebo-controlled, multicenter, polysomnographic study of gabapentin in transient insomnia induced by sleep phase advance. J Clin Sleep Med. 2014 Oct 15;10(10):1093-100. doi: 10.5664/jcsm.4108. PMID 25317090
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451157&StudyName=A%20Polysomnographic%20Study%20Of%20Single-Dose%20Gabapentin%20In%20Transient%20Insomnia%20